CLINICAL TRIAL: NCT01107704
Title: A Randomized Controlled Trial to Test the Effectiveness of a Multi-faceted Communication Intervention for Family Members of Critically Ill Patients.
Brief Title: Family Support Intervention in Intensive Care Units (The Four Supports Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K23AG032875 (NIH); K23AG032875 (NIH)
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Physician-Family Communication in Intensive Care Units; Surrogate Decision-making for Critically Ill Patients
Keywords: Intensive Care Units; Surrogates; Family Members; Physicians; Critically Ill; Depression; Anxiety; Emotional; Support; Multi-faceted communication; Grief; Prognosis; Family Support Counselor
MeSH Terms: conditions — Critical Illness; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Support Intervention (Experimental)
  Interventions: Behavioral: Family Support Intervention
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Family Support Intervention — Multifaceted family support intervention
  Arms: Family Support Intervention

SUMMARY:
The purpose of this study is to test the effectiveness of a multi-faceted communication intervention for family members of critically ill patients to reduce the family members' long-term symptoms of depression and anxiety.

DETAILED DESCRIPTION:
One in four elderly Americans die in or shortly after discharge from an intensive care unit. An expanding body of literature documents that physician-family communication and end-of-life care is poor in intensive care units. These deficiencies are associated with high rates of adverse psychological outcomes among surrogates, physician-family conflict, and life support decisions that may be inconsistent with patients' goals and preferences. There is a lack on information on practical, generalizable interventions that effectively improve this important aspect of care for elderly patients and their families.

The primary aim of this study is to evaluate the effectiveness of a multifaceted communication intervention to improve psychological outcomes among family members of critically ill patients, using a randomized, controlled trial design.

ELIGIBILITY:
Inclusion Criteria for ICU Patients:

* must be unable to make treatment decisions for him/herself, as determined by the patient's physicians.
* must have have either an APACHE II score of ≥ 25 or, for patients with a primary neurologic diagnosis (e.g. intracranial hemorrhage, subdural hemorrhage, or subarachnoid hemorrhage), physician estimate that the patient has at least a 50% risk of long term, severe functional impairment
* must be 50 years old or greater.

Exclusion Criteria for ICU Patients:

* Patients who do not have surrogates or at least one family member who is willing to participate in the study.
* Patients awaiting organ transplantation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2010-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Family Outcome: Family members' depressive symptoms | Three months following patient death or discharge from the ICU.
Patient Outcome: Patient centeredness of care | Three months following patient death or discharge from the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B. White, MD, MAS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania, United States